CLINICAL TRIAL: NCT00118950
Title: Effect of Metformin Versus Repaglinide Treatment on Glycemic Control and Non-Glycaemic Cardiovascular Risk Factors in Non-Obese Type 2 Diabetic Patients Uncontrolled by Diet
Brief Title: Effect of Metformin Versus Repaglinide Treatment in Non-Obese Type 2 Diabetic Patients Uncontrolled by Diet
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ReMet
Record Dates: First submitted 2005-07-01; First posted 2005-07-12 (Estimated); Last update posted 2008-12-08 (Estimated); Status verified 2008-12

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; repaglinide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 4 (Active Comparator): Metformin plus placebo-Repgalinide. Double-masked, randomized. Duration: Four months.
  Interventions: Drug: Metformin; Drug: Placebo-Repaglinide.
- 2 (Active Comparator): Repaglinide plus Placebo-Metformin. Double-masked, randomized. Duration: Four months.
  Interventions: Drug: Repaglinide; Drug: Placebo-Metformin.
- 1 (Other): Run-in period: Treatment: Diet-only. Duration: One month.
  Interventions: Other: Diet-only.
- 3 (Other): Wash-out period: Treatment: Diet-only: Duration: One month.
  Interventions: Other: Diet-only.

INTERVENTIONS:
Drug: Metformin — Tablet Metformin 500 mg; Dosage: 1000 mg two times daily. Duration: Four months.
  Arms: 4
Drug: Repaglinide — Tablet Repaglinide 1 mg; Dosage: 2 mg three times daily. Duration: Four months.
  Arms: 2
Drug: Placebo-Metformin. — Tablet Placebo (corresponding to 500 mg Metformin). Dosage: 2 tablets two times daily. Duration: Four months.
  Arms: 2
Drug: Placebo-Repaglinide. — Tablet Placebo (corresponding to 1 mg Repaglinide). Dosage: 2 tablets three times daily. Duration: Four months.
  Arms: 4
Other: Diet-only. — Diet-only treatment. Duration: One month.
  Arms: 1; 3

SUMMARY:
Background: Metformin is the first drug of choice in obese patients with type-2 diabetes (T2DM) due to its antiglycaemic as well as its cardiovascular protective potentials. In non-obese T2DM patients insulin-secretagogues are empirically used as first choice. The aim of this study was to evaluate the effect of metformin versus an insulin-secretagogue, repaglinide on glycaemic regulation and non-glycaemic cardiovascular risk markers in non-obese patients with T2DM.

Methods: Single-center, randomised, double-masked, double-dummy, cross-over-study of 96 non-obese (BMI ≤ 27 kg/m2) Caucasian T2DM-patients. After a one month run-in on diet-only treatment, patients were randomised to either repaglinide 2mg three times a day (t.i.d). followed by metformin 1g twice a day (b.i.d.) or vice versa each for a period of four months with a one month wash-out between interventions.

ELIGIBILITY:
Inclusion Criteria:

Type-2 diabetes, defined as:

* Age at onset of diabetes ≥ 40 years
* Fasting serum C-peptide ≥ 300 pmol/l or a non-fasting or glucagon-stimulated serum C-peptide ≥ 600 pmol/l
* No history of ketonuria or ketoacidosis.
* BMI ≤ 27 kg/m2.
* Fasting plasma-glucose ≥ 6.5 mmol/l after at least one month of diet-only treatment.
* HbA1c ≤ 9.5% at ongoing oral anti-hyperglycaemic agents. HbA1c ≥ 6.5% after minimum one month of diet-only treatment.
* Weight-loss of no more than 5.0 kg during the last 6 months prior to enrolment.

Exclusion Criteria:

* Type-1 diabetes
* Insulin-treated type-2 diabetes
* Secondary diabetes, heart-failure
* Serum-creatinine above the upper limit
* Serum-ASAT elevated more than 3 fold above the upper limit
* Factor II-VII-X decreased below 0.7
* Ongoing coexisting illnesses with a life-shortening prognosis
* Mental retardation or reduced intellectual behaviour
* Pregnancy
* History of drug-abuse or HbA1c>10.5% at two separate visits with at least one month interval during treatment-periods.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-03; Study Completion 2003-03

PRIMARY OUTCOMES:
HaemoglobinA1c

SECONDARY OUTCOMES:
Home-monitored 7-point plasma-glucose profiles
Body-weight
Waist- and hip-circumference
Fasting and postprandial (after a standard test-meal) measures of plasma-glucose, insulin, c-peptide, free fatty acids, lipoproteins, triglycerides and other markers related to lipid-metabolism (e.g. apo-lipoproteins, lipoprotein particle size etc.).
Biomarkers related to inflammation, endothelial dysfunction and fibrinolysis (e.g. hs-CRP, TNF-alpha, IL-6, ICAM, VCAM, E-selectin, vWF, PAI-1 and t-PA, adiponectin, ADMA, AGE-peptides).
Albuminuria and 24-hour blood-pressure measurements.
Platelet aggregation, markers of platelet activity and fibrinolytic markers fasting as well as before and after physical activity.
DNA for genotyping.
Adverse events and safety variables (e.g. hypoglycaemia, haemoglobin, white blood cell count, cobalamine and folate).

CONTACTS AND LOCATIONS:
Overall Officials: Allan A Vaag, M. D., Chief Physician, Study Chair — Steno Diabetes Center Copenhagen; Soeren S Lund, M. D., Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center, Gentofte Municipality, Denmark